CLINICAL TRIAL: NCT05049616
Title: Oral Combined Hydrochlorothiazide/Lisinopril Versus Oral Nifedipine for Postpartum Hypertension: A Comparative Effectiveness Pilot Randomized Controlled Trial
Brief Title: Oral Combined Hydrochlorothiazide/Lisinopril Versus Oral Nifedipine for Postpartum Hypertension
Acronym: ACE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Michal Fishel Bartal, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-21-0476
Record Dates: First submitted 2021-08-31; First posted 2021-09-20 (Actual); Results first posted 2023-08-14 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Hypertension in Pregnancy; Postpartum Preeclampsia
MeSH Terms: conditions — Hypertension, Pregnancy-Induced | interventions — Angiotensin-Converting Enzyme Inhibitors; Diuretics

STUDY DESIGN:
Intervention Model Description: randomized control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hctz/Lisinopril (Experimental): Hctz/Lisinopril for postpartum management of hypertension. either a combined pill of ACE inhibitors and diuretics (Hydrochlorothiazide/Lisinopril)
  Interventions: Drug: ACE Inhibitors and Diuretics
- Extended release nifedipine (Active Comparator): calcium channel blocker (Nifedipine
  Interventions: Drug: NIFEdipine ER

INTERVENTIONS:
Drug: ACE Inhibitors and Diuretics — Hctz/Lisinopril (brand name: Zestoretic)
  Arms: Hctz/Lisinopril
Drug: NIFEdipine ER — Extended release nifedipine
  Arms: Extended release nifedipine

SUMMARY:
The purpose of this study is to see if a combined pill of Angiotensin-converting enzyme (ACE) inhibitors (a medication that helps relax your veins and arteries to lower your blood pressure) with diuretics (sometimes called water pills, help rid your body of salt and water) will control blood pressure better than a different blood pressure medication of calcium channel blocker (lower your blood pressure by preventing calcium from entering the cells of your heart and arteries). Both medications are part of our usual care for high blood pressure after delivery.

DETAILED DESCRIPTION:
In individuals with preeclampsia, persistent hypertension and edema result in part from the mobilization of up to 8 liters of fluid and sodium from the extravascular to intravascular space. The increased urinary sodium excretion on days 3-5 postpartum likely results from higher atrial natriuretic peptide concentrations in plasma and activation of the renin-angiotensin-aldosterone system. Adding diuretics for postpartum hypertension has been associated with better blood pressure control in some of the studies.

* CVD is the leading cause for mortality worldwide.
* Primary prevention is more effective than treating CVD.
* Pregnancy is often the 1st adult engagement with the healthcare system.
* Preeclampsia is a risk factor for long term CVD, even after controlling for mutual risk factors.
* CVD is the leading cause for pregnancy related mortality.
* There is no good data regarding the optimal medications to control blood pressure after delivery.
* ACE inhibitors play an important role in controlling blood pressure outside of pregnancy and there is extensive evidence to support their cardioprotective effects.
* The optimal use of diuretics in the postpartum in patients with preeclampsia, require further study and clarification to augment current management schemes.

Hypothesis: that in postpartum women with hypertensive disorders, oral combined Hydrochlorothiazide/Lisinopril will reduce postpartum hypertension at 7 days after delivery compared to usual care with calcium channel blockers.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum women at ≥ 18 years of age
* Postpartum diagnosis of persistent hypertension (2 measurements of Systolic BP ≥150 and/or diastolic BP ≥ 100 or systolic BP ≥140 and/or diastolic BP ≥ 90 for people with diabetes) requiring an oral medication based on the ACOG criteria or
* Hypertensive disorder of pregnancy diagnosed antepartum or intrapartum requiring blood pressure medication in the postpartum
* Chronic hypertension requiring blood pressure medication postpartum

Exclusion Criteria:

* Urine output < 30 cc/h prior to screening for eligibility
* Creatinine > 1.4 during current admission
* End-stage renal disease
* Hypersensitivity to ACE inhibitors or sulfa drugs
* Idiopathic/hereditary angioedema
* Hyperkalemia (serum potassium >5 mEq/L) during current admission
* Pulmonary edema

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2022-06-26 (Actual); Study Completion 2023-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michal Fishel Bartal, MD, Principal Investigator — UT Health Science Center
Locations (1):
- University of Texas Health Science Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hctz/Lisinopril | Extended release nifedipine
Started | 34 | 36
Completed | 31 | 36
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hctz/Lisinopril | Extended release nifedipine | Total
Number analyzed (Participants) | 31 | 36 | 67
Age, Customized [Count of Participants; unit: Participants]
  <35 years | 24 | 20 | 44
  >=35 years | 7 | 16 | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 36 | 67
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 3 | 4 | 7
  Non-Hispanic Black | 16 | 24 | 40
  Hispanic | 9 | 7 | 16
  Asian | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 31 | 36 | 67
Number of participants with private insurance for prenatal care [Count of Participants; unit: Participants] | 7 | 18 | 25
Number of participants that are Married/living with partner [Count of Participants; unit: Participants] | 11 | 14 | 25
Number of participants with Nulliparous [Count of Participants; unit: Participants] | 4 | 7 | 11
Pre-pregnancy Body Mass Index [Median (Inter-Quartile Range); unit: kg/m^2] | 40.1 [33.8 to 46.3] | 37.8 [34.6 to 43.4] | 38.5 [35.1 to 43.4]
Number of participants with a BMI ≥ 30 [Count of Participants; unit: Participants] | 20 | 25 | 45
Number of participants with Diabetes diagnosed prior to pregnancy [Count of Participants; unit: Participants] | 6 | 7 | 13
Number of participants with Gestational diabetes [Count of Participants; unit: Participants] | 2 | 5 | 7
Number of participants with Thyroid disease [Count of Participants; unit: Participants] | 1 | 3 | 4
Number of participants who Smoke during pregnancy [Count of Participants; unit: Participants] | 1 | 4 | 5
Number of participants with Alcohol use during pregnancy [Count of Participants; unit: Participants] | 0 | 1 | 1
Number of participants with Substance use during pregnancy [Count of Participants; unit: Participants] | 1 | 5 | 6
Number of participants with Chronic hypertension [Count of Participants; unit: Participants] | 14 | 15 | 29
Number of participants who Use Blood Pressure medication during pregnancy [Count of Participants; unit: Participants] | 15 | 13 | 28
Number of participants with Hypertensive disorder during pregnancy [Count of Participants; unit: Participants] — Hypertensive disorder including gestational hypertension, preeclampsia, or superimposed preeclampsia.
  Participants | 28 | 31 | 59
Number of participants with Preeclampsia with severe features [Count of Participants; unit: Participants] | 24 | 27 | 51
Number of participants with New onset postpartum hypertension [Count of Participants; unit: Participants] | 0 | 5 | 5
Number of participants who had labor induced [Count of Participants; unit: Participants] | 9 | 18 | 27
Gestational weeks at delivery [Median (Inter-Quartile Range); unit: weeks] | 34.4 [31.9 to 36.7] | 36.6 [35.1 to 37.7] | 35.4 [34.2 to 36.5]
Number of pre-term delivery [Count of Participants; unit: Participants] | 25 | 20 | 45
Number of Cesarean delivery [Count of Participants; unit: Participants] | 23 | 20 | 43
Number of participants who Need IV Blood Pressure medications prior to randomization [Count of Participants; unit: Participants] | 11 | 11 | 22
Postpartum day at randomization [Median (Inter-Quartile Range); unit: days] | 1.4 [0.9 to 1.8] | 1.0 [0.6 to 2.2] | 1.2 [0.8 to 1.9]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Stage 2 Hypertension
Description: Stage 2 hypertension at day 7-10 after delivery (defined as SBP ≥ 140 and/or DBP ≥ 90 mmHg) or admission to the hospital for blood pressure control prior to day 10.
  Primary outcome will be calculated as the average BP reading for day 7-10 after delivery.
Time Frame: 7-10 after delivery
Population: Data were not collected for 1 participants in the Hctz/Lisionpril arm. Data were not collected for 8 participants in the extended release nifedipine arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Hctz/Lisinopril | Extended release nifedipine
Number analyzed (Participants) | 30 | 28
Participants | 8 | 12

2. Secondary Outcome: Number of Participants With Severe Postpartum Hypertension
Description: severe postpartum hypertension (SBP≥160 and/or DBP≥110 mmHg on 2 occasions, 15 minutes apart)
Time Frame: 7-10 after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Hctz/Lisinopril | Extended release nifedipine
Number analyzed (Participants) | 31 | 36
Participants | 6 | 5

3. Secondary Outcome: Number of Participants Who Received Additional Antihypertensive During Admission
Description: number of participants who received additional antihypertensive during admission, at 7-10 days postpartum.
Time Frame: 7-10 days postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Hctz/Lisinopril | Extended release nifedipine
Number analyzed (Participants) | 31 | 36
Participants | 6 | 5

4. Secondary Outcome: Postpartum Length of Stay
Description: time spent in hospital following delivery
Time Frame: up to 30 days after delivery
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Hctz/Lisinopril | Extended release nifedipine
Number analyzed (Participants) | 31 | 36
days | 4 [3 to 5] | 3 [3 to 4]

5. Secondary Outcome: Postpartum Readmission
Description: occurrence of returning to hospital for admission postpartum
Time Frame: up to 30 days after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Hctz/Lisinopril | Extended release nifedipine
Number analyzed (Participants) | 31 | 36
Participants | 5 | 1

6. Secondary Outcome: Time to Blood Pressure Control
Description: The time from delivery to Blood Pressure control (i.e time from delivery to last BP <150/100).
Time Frame: 10 days
Population: Data were not collected for this outcome measure.
Arm/Group | Hctz/Lisinopril | Extended release nifedipine
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Incidence of Persistent Postpartum Hypertension
Description: Incidence of persistent postpartum hypertension 6 weeks postpartum (SBP ≥ 140 and/or DBP ≥ 90 mmHg).
Time Frame: 6 weeks postpartum
Population: Data were not collected for this outcome measure.
Arm/Group | Hctz/Lisinopril | Extended release nifedipine
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Occurrence of Proteinuria
Description: Proteinuria is measured by urine protein creatinine ratio
Time Frame: 7-10 days, and 6 weeks postpartum
Population: Data were not collected for this outcome measure
Arm/Group | Hctz/Lisinopril | Extended release nifedipine
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Presense of Labs Abnormality
Description: Labs abnormality including hyperkalemia or creatinine increase
Time Frame: 7-10 days, and 6 weeks postpartum
Population: Data were not collected for this outcome measure
Arm/Group | Hctz/Lisinopril | Extended release nifedipine
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Compliance With Medications
Description: Compliance with medications. The patient will be asked to bring their medication bottle with them and the compliance will be measured by counting pills at each postpartum visit.
Time Frame: at the time of the 1st postpartum clinic visit, which is about 6 to 37 days after birth
Population: Data were not collected for 4 participants in the Hctz/Lisinopril arm. Data were not collected for 8 participants in the Extended release nifedipine arm
Measure: Count of Participants; unit: Participants
Arm/Group | Hctz/Lisinopril | Extended release nifedipine
Number analyzed (Participants) | 27 | 28
Participants | 22 | 26

11. Secondary Outcome: Time to Control Blood Pressure
Description: Blood pressure at 3 month, 6 month, 9 month, 1 year after delivery and need for BP medications. Definition of controlled blood pressure is (SBP < 140 and/or DBP < 90 mmHg). This will be assessed by telephone encounter with the patient
Time Frame: 3 month-1 year
Population: Data were not collected for this outcome measure.
Arm/Group | Hctz/Lisinopril | Extended release nifedipine
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Number of Patients Receiving Primary Care With BP Measurement
Description: Number of patients receiving primary care with BP measurement at 1 year
Time Frame: 1 year postpartum
Population: Data were not collected for this outcome because participants were lost to follow up.
Arm/Group | Hctz/Lisinopril | Extended release nifedipine
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Postpartum Complications- Number of Participants With ICU Admission
Description: Need for ICU admission
Time Frame: 10 days postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Hctz/Lisinopril | Extended release nifedipine
Number analyzed (Participants) | 31 | 36
Participants | 2 | 0

14. Secondary Outcome: Postpartum Complications- Number of Participants With HELLP (Hemolysis, Elevated Liver Enzymes and Low Platelets) Syndrome
Description: Hemolysis, elevated liver enzymes, low platelet count: HELLP
Time Frame: 10 days postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Hctz/Lisinopril | Extended release nifedipine
Number analyzed (Participants) | 31 | 36
Participants | 1 | 0

15. Secondary Outcome: Postpartum Complications- Number of Participants With Eclampsia
Description: Eclampsia, which is considered a complication of severe preeclampsia, is commonly defined as new onset of grand mal seizure activity and/or unexplained coma during pregnancy or postpartum in a woman with signs or symptoms of preeclampsia.
Time Frame: 10 days postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Hctz/Lisinopril | Extended release nifedipine
Number analyzed (Participants) | 31 | 36
Participants | 0 | 0

16. Secondary Outcome: Postpartum Complications- Number of Participants With Stroke
Description: Stroke
Time Frame: 10 days postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Hctz/Lisinopril | Extended release nifedipine
Number analyzed (Participants) | 31 | 36
Participants | 0 | 0

17. Secondary Outcome: Postpartum Complications- Number of Participants With Renal Failure
Description: Renal failure
Time Frame: 10 days postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Hctz/Lisinopril | Extended release nifedipine
Number analyzed (Participants) | 31 | 36
Participants | 0 | 0

18. Secondary Outcome: Postpartum Complications- Number of Participants With Pulmonary Edema
Description: Pulmonary edema
Time Frame: 10 days postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Hctz/Lisinopril | Extended release nifedipine
Number analyzed (Participants) | 31 | 36
Participants | 1 | 0

19. Secondary Outcome: Postpartum Complications - Number of Participants With Cardiomyopathy
Description: Cardiomyopathy
Time Frame: 10 days postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Hctz/Lisinopril | Extended release nifedipine
Number analyzed (Participants) | 31 | 36
Participants | 1 | 0

20. Secondary Outcome: Postpartum Complications- Number of Participants With Maternal Death
Description: Maternal death
Time Frame: 10 days postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Hctz/Lisinopril | Extended release nifedipine
Number analyzed (Participants) | 31 | 36
Participants | 0 | 0

21. Secondary Outcome: Receipt of Additional Antihypertensive During Admission
Description: Receipt of additional antihypertensive during admission at 6 weeks postpartum
Time Frame: 6 weeks postpartum
Population: Data were not collected for this outcome measure
Arm/Group | Hctz/Lisinopril | Extended release nifedipine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 6 weeks post delivery
Arm/Group | Hctz/Lisinopril | Extended release nifedipine
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/36
Serious Adverse Events (participants affected / at risk) | 2/34 | 0/36
Other Adverse Events (participants affected / at risk) | 0/34 | 0/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hctz/Lisinopril (N=34) | Extended release nifedipine (N=36)
Intensive care unit admission (General disorders) | 2 | 0
HELLP (Hemolysis, Elevated Liver enzymes and Low Platelets) syndrome (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-06): https://cdn.clinicaltrials.gov/large-docs/16/NCT05049616/Prot_SAP_000.pdf